CLINICAL TRIAL: NCT03878251
Title: Development and Validation of Quantitative Attention Evaluation Criteria in Patients With Intellectual Disability
Brief Title: Outcomes Measures in Intellectual Disability
Acronym: EVALDI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Plateforme PRISME (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: K180106J; 2018-A00686-49 (Registry Identifier: IDRCB)
Record Dates: First submitted 2019-03-14; First posted 2019-03-18 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Attention Deficit in Intellectual Disability
Keywords: Intellectual disability; Attention evaluation criteria; Games on touchscreen; Eye tracking
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- X fragile syndrome patients (Other)
  Interventions: Device: Quantitative attention evaluation criteria in intellectual disability
- Angelman syndrome patients (Other)
  Interventions: Device: Quantitative attention evaluation criteria in intellectual disability
- Rett syndrome patients (Other)
  Interventions: Device: Quantitative attention evaluation criteria in intellectual disability
- Patients with other genetic rare syndromes with intellectual d (Other)
  Interventions: Device: Quantitative attention evaluation criteria in intellectual disability

INTERVENTIONS:
Device: Quantitative attention evaluation criteria in intellectual disability — Quantitative interactive attention evaluation tests by using games on touchscreen and or eye tracking (oculometer)

SUMMARY:
Objective quantitative primary endpoints are lacking in Clinical trials in intellectual disability. We propose to develop quantitative interactive attention evaluation criteria in patients with intellectual disability by using games on touchscreen and or eye tracking.

DETAILED DESCRIPTION:
The aim of the study is to develop and validate quantitative interactive attention evaluation criteria by using games on touchscreen and or eye tracking in patients with intellectual disability. Tests will have to be suitable whatever severity and etiology of intellectual disability. Tests have to evaluate attention and concentration troubles in intellectual disability.Once validated, tests could be used as outcome measures in clinical trials and as cognitive reeducation tools in intellectual disability.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both sex, with intellectual disability
2. Minor patients 6 years old or more (age corresponding to the end of regression period observed in Rett patients) or major protected patients
3. Patients with more or less severe intellectual disability from various causes including Fragile X syndrome, Rett syndrome, Angelman syndrome and other etiologies of intellectual disabilities and intellectual disabilities without identified etiology
4. Affiliation to a social security system own or affiliated (excluding AME)
5. Presence of parents or legal representative
6. Informed consent signed by parents or legal representative

Exclusion Criteria:

1. Behavioral disorders not compatible with interactive tool (major agitation, straight and self aggressiveness)
2. Uncontrolled seizure disorder despite treatment

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2022-06-07 (Actual); Study Completion 2022-06-07 (Actual)

PRIMARY OUTCOMES:
Correlation between number of successful attempts and intellectual disability evaluated by Intelligence quotient (IQ) or age of development | up to 3 months
  Test performed 1 time during a visit (1 day) can be repeated (for a maximum of 15 patients) within 3 months if an adaptation of the interactive tool is necessary

SECONDARY OUTCOMES:
Maximal reached level for each test | up to 3 months
Number of errors during the test | up to 3 months
Time to reach each level of the test | up to 3 months
Time to reach maximum level of the test | up to 3 months
Total test duration | up to 3 months
Fixing time for eye tracking | up to 3 months
Successful test numbers in each level | up to 3 months
Correlation with Intelligence quotient (IQ) or age of development according to intellectual disability severity | up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: CHARLES Perrine, MD PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital La Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No